CLINICAL TRIAL: NCT02320643
Title: A Prospective Pilot Study to Investigate the Efficacy of Partially Absorbable Mesh(Seratom PA®) in Patients With Pelvic Organ Prolapsed
Brief Title: A Pilot Study to Investigate the Efficacy of Partially Absorbable Mesh in Patients With Pelvic Organ Prolapsed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POP-SERATOM PA
Record Dates: First submitted 2014-12-09; First posted 2014-12-19 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Pelvic Organ Prolapse
Keywords: Partially absorbable mesh
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Seratom® PA mesh (Experimental): Partially absorbable mesh
  Interventions: Device: Seratom® PA mesh

INTERVENTIONS:
Device: Seratom® PA mesh — Partially absorbable mesh

SUMMARY:
The purpose of this study is to evaluate the efficacy, recurrence, postoperative complications of partially absorbable mesh(Seratom®PA) in patients with pelvic organ prolapse.

DETAILED DESCRIPTION:
Patients with pelvic organ prolapse are administrated partially absorbable mesh(Seratom®PA). It is performed pelvic organ prolapse quantification(POP-Q) examination, quality of life(QOL) questionnaire complications at postop 2week, 12week, 24week.

ELIGIBILITY:
Inclusion Criteria:

1. Woman who aged 41 years or older
2. Subjects who have symptomatic pelvic organ prolapse quantification(POP-Q) stage II & cystocele or higher requiring surgical repair
3. Subjects who desires vaginal reconstructive surgery
4. Subjects who have uterus < 12 weeks size
5. Subjects who are able to complete study questionnaires and assessment
6. Subjects who are available for 6 months follow-up

Exclusion Criteria:

1. Subjects who have medical contractions, e.g. current urinary tract, vaginal or pelvic infection, history of pelvic irradiation, history of lower urinary tract malignancy, chronic steroid use, or a compromised immune system
2. Subjects who have received anticoagulation therapy
3. Subjects who are on current intermittent catheterization
4. Subjects whose BMI is over 30kg/m2
5. Subjects who have uncontrolled diabetes
6. Subjects who are on any medication which could result in compromised immune response, such as immune modulators
7. Subjects who are currently pregnant or intends to become pregnant during the study period or <12 months post-partum
8. Subjects who have received other laparoscopic or abdominal or pelvic surgery in the past 1 months
9. Subjects who need for concomitant surgery requiring an abdominal incision
10. Subjects who have had a prior prolapse implant procedure (i.e. IVS tunneler, Perigee, Apogee, graft augmented repair, etc)

    * Note: previous traditional repairs are allowed.
11. Subjects who have had radiation therapy to the pelvic area
12. Subjects who have pelvic cancer or have had pelvic cancer within the past 12 months or have had on cytostatic medication within the past 12 months
13. Subjects who have a shortened vagina or other known Mullerian anomaly (e.g. uterine didelphys.)
14. Subjects who have a known neurologic or medical condition affecting bladder function (e.g. Multiple Sclerosis, spinal cord injury)
15. Subjects who have a known hypersensitivity to the graft material(s)

Min Age: 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse Quantification(POP-Q) stage | Change from baseline in Pelvic Organ Prolapse Quantification(POP-Q) stage at postop 2week, 12week, 24week
Surgical revision rate | For post op 6 months from baseline

SECONDARY OUTCOMES:
No of patients complications occurred | For post op 6 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kwon Sang Hoon, Doctor, Principal Investigator — Keimyung University Dongsan Medical Center
Locations (1):
- Samyang Biopharmaceuticals, Seoul, South Korea